CLINICAL TRIAL: NCT02903459
Title: Analyze the Relationship Between the Density of Abdominal Visceral and Subcutaneous Fat and Cellulite With the Lumbar
Brief Title: Analyze the Relationship Between the Density of Fat Tissue and Cellulite With the Lumbar Lordosis Degree
Status: Completed | Type: Observational
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Andreia Noites, Professor, Escola Superior de Tecnologia da Saúde do Porto
Other Study IDs: AN-005; AR (Other: Escola Superior de Tecnologia da Saúde do Porto); MS (Other: Escola Superior de Tecnologia da Saúde do Porto); MC (Other: Escola Superior de Tecnologia da Saúde do Porto)
Record Dates: First submitted 2016-08-01; First posted 2016-09-16 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Lordosis
Keywords: Central Fat; Subcutaneous Fat; Lumbar Lordosis Degree; Cellulite
MeSH Terms: conditions — Lordosis; Cellulite

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Males: Evaluation of body mass index, determination of waist-to-hip ration and waist-to-height ration, using perimetry; evaluation of 7 skinfold according to the model 7-site-skinfold Equation, by Jackson and Pollock, and photogrammetry (to evaluate the lumbar lordosis degree) in males aged between 18 and 26.
  Interventions: Other: Transversal Study so there is no intervention
- Young Adults: Evaluation of abdominal thickness, percentage of abdominal fat and photogrammetry (to evaluate the lumbar lordosis degree) in young adults females aged between 18-26.
  Interventions: Other: Transversal Study so there is no intervention
- Adults: Evaluation of abdominal thickness, percentage of abdominal fat and photogrammetry (to evaluate the lumbar lordosis degree) in adult females aged between 40-60.
  Interventions: Other: Transversal Study so there is no intervention
- Females: Evaluation of body mass index, determination of waist-to-hip ration and waist-to-height ration using perimetry, evaluation of 7 skinfold according to the model 7-site-skinfold Equation, by Jackson and Pollock, and photogrammetry (to evaluate the lumbar lordosis degree) in females aged between 18 and 26.
  Interventions: Other: Transversal Study so there is no intervention

INTERVENTIONS:
Other: Transversal Study so there is no intervention

SUMMARY:
The aim of this study is analyze the relationship between the density of visceral and subcutaneous fat and cellulite with the lumbar lordosis degree.

DETAILED DESCRIPTION:
There are two types of abdominal fat: subcutaneous adipose tissue which is more superficial, lying above the abdominal muscle wall and visceral adipose tissue, corresponding to the intra-abdominal fat witch is more harmful to health.

The accumulation of fat tissue differs between genders and age. Men have a huge propensity for developing central fat and women accumulate more subcutaneous fat tissue on the gluteal-femoral region. Some authors suggest that the accumulation of fat tissue increases with age.

Several studies have concluded that there is a relationship between the abdominal fat storage and the degree of lumbar curvature.

In addition, some authors also suggest that there is a relationship between the degree of lumbar lordosis and cellulite, which is related to circulatory changes.

However these relationships are not yet clarified in the literature.

ELIGIBILITY:
Inclusion Criteria: All the community of the School of Allied Health Technologies; aged between 18-60

Exclusion Criteria: Pathologies (cardiovascular, metabolic, cancer, respiratory, muscular); pregnancy; abdominoplasty; collum and gluteal surgeries; deregulated menstrual cycle ; anatomical changes; anticelulitic treatments

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All the comunity of the School of Allied Health Technologies
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-06; Primary Completion 2016-10 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of Lumbar Lordosis by analysing photos of the lateral right side of the participants | Day 1
  We used photogrammetry for this evaluation. We marked the anatomical points (T11, L1, S2 and Antero-superior Iliac Spine) with isopod balls. We took a picture of the right lateral view of the participant. Finally we used the SAPo software to measure free angles to determinate lumbar lordosis degree.

SECONDARY OUTCOMES:
Body Mass Index | Day 1
  The height was measured by a tape-measure. We used the bioimpedance balance to determinate the body mass of the participants. BMI was calculated by using the body weight divided by height squared.
Perimeters measurements using a tape-measure at waist level and at trochanters level at the end of expiration | Day 1
  The perimeters measurements were done at the end of expiration, at waist level and at trochanters level. The waist-hip ratio was calculated by using the waist level perimeter divided by trochanters level perimeter and the waist-to-height ratio was calculated by using the waist level perimeter divided by height
Skinfold measures | Day 1
  Subscapular, tricipital, chest, axillar, suprailiac, abdominal, thick skinfolds were performed three times in right hemibody, by caliper according to the model 7-site-skinfold Equation, by Jackson and Pollock. Siri equation was used to determinate the percentage of total body fat.
Bioimpedance Balance | Day 1
  This instrument was used to determine the weight, the percentage of body and abdominal fat, the visceral index and the percentage of body and abdominal lean mass.
Ecograph | Day 1
  It was used for distinguishing of abdominal thickness fat (differentiate the fat in visceral and subcutaneous fat tissue) and in order to obtain the thickness of the subcutaneous adipose tissue at the points of maximum and minimum temperature on the gluteal region.
Thermography | Day 1
  Measurement of skin temperature in the gluteal region to obtain the average, the minimum and the maximum temperature on this area.
Cellulite Grading Scale | Day 1
  6 Photos were taken in the posterior and lateral (right and left) views, 3 in relaxation and 3 in gluteal isometric contraction.

OTHER OUTCOMES:
International Physical Activity Questionnaire | Day 1
  International Physical Activity Questionnaire was used to monitor lifestyle
Food Frequency Questionnaire | Day 1
  Food Frequency Questionnaire was used to monitor lifestyle

CONTACTS AND LOCATIONS:
Overall Officials: Andreia Noites, PhD, Principal Investigator — Escola Superior de Tecnologia da Saúde do Porto
Locations (1):
- Andreia Noites, Vila Nova de Gaia, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jackson AS, Pollock ML. Generalized equations for predicting body density of men. Br J Nutr. 1978 Nov;40(3):497-504. doi: 10.1079/bjn19780152. PMID 718832
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Siqueira, G. R., Alencar, G. G., Rocha, M. B. N., Silva, L. R., Moura, M. C. G. G., & Silva, G. A. P. (2015). Relação entre lordose lombar e depósito de gordura abdominal em adolescentes e adultos jovens. Revista Brasileira de Ciência e Movimento, 74-80.
- [Background] Power ML, Schulkin J. Sex differences in fat storage, fat metabolism, and the health risks from obesity: possible evolutionary origins. Br J Nutr. 2008 May;99(5):931-40. doi: 10.1017/S0007114507853347. Epub 2007 Nov 1. PMID 17977473
- [Background] Lopes C, Aro A, Azevedo A, Ramos E, Barros H. Intake and adipose tissue composition of fatty acids and risk of myocardial infarction in a male Portuguese community sample. J Am Diet Assoc. 2007 Feb;107(2):276-86. doi: 10.1016/j.jada.2006.11.008. PMID 17258965
- [Background] Kuo YL, Tully EA, Galea MP. Video analysis of sagittal spinal posture in healthy young and older adults. J Manipulative Physiol Ther. 2009 Mar-Apr;32(3):210-5. doi: 10.1016/j.jmpt.2009.02.002. PMID 19362231
- [Background] Bazzocchi A, Filonzi G, Ponti F, Sassi C, Salizzoni E, Battista G, Canini R. Accuracy, reproducibility and repeatability of ultrasonography in the assessment of abdominal adiposity. Acad Radiol. 2011 Sep;18(9):1133-43. doi: 10.1016/j.acra.2011.04.014. Epub 2011 Jul 2. PMID 21724427
- [Background] Noites A, Nunes R, Gouveia AI, Mota A, Melo C, Viera A, Adubeiro N, Bastos JM. Effects of aerobic exercise associated with abdominal microcurrent: a preliminary study. J Altern Complement Med. 2015 Apr;21(4):229-36. doi: 10.1089/acm.2014.0114. PMID 25875939
- [Background] Nkengne A, Papillon A, Bertin C. Evaluation of the cellulite using a thermal infra-red camera. Skin Res Technol. 2013 Feb;19(1):e231-7. doi: 10.1111/j.1600-0846.2012.00633.x. Epub 2012 Jun 29. PMID 22741614
- [Background] Goldman, M., & Hexsel, D. (2006). Cellulite: Pathophysiology and Treatment (i. healthcare Ed. 2ª edição ed.).
- [Background] FLIR. (2013). Flir E-Series.
- [Background] COMED. (2013). Company Comed.
- [Background] Corporation, T. (2006). Tanita: Monitoring Your Heath. Tanita Manual: InnerScan Body Composition Monitor